CLINICAL TRIAL: NCT06296511
Title: The Influence of Acute Moderate-intensity Continuous Exercise on Appetite Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Professor David Stensel, Professor, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Loughborough University
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Obesity; Overweight
Keywords: Exercise; Appetite; Oxyntomodulin; Growth differentiation factor 15; GDF-15
MeSH Terms: conditions — Obesity; Overweight; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Participants were asked to arrive at the lab at 8.30 am, having fasted overnight for 10 hours. After resting in the lab for 30 minutes, participants were asked to exercise at an intensity of 70 percent of their peak oxygen uptake for an hour before resting in the lab for a further 2.5 hours. Ad libitum energy intake was assessed 1 h after exercise completion.
  Interventions: Behavioral: Exercise
- Control (No Intervention): Participants replicated all the procedures of the exercise trial except they rested for 1 h as the exercise counterpart.

INTERVENTIONS:
Behavioral: Exercise — 60 min of treadmill exercise performed at 70% of peak oxygen uptake.
  Arms: Exercise

SUMMARY:
A key area of obesity research has focused on the link between appetite, energy balance and weight control. Within this area, several appetite-related hormones and cellular cytokines have been identified as key signals influencing appetite and food intake. This includes the appetite-suppressing hormone oxyntomodulin (OXM) and a cellular stress-induced cytokine growth differentiation factor 15 (GDF-15).

The aims of this study are: (1) to investigate the effect of acute moderate-intensity continuous exercise on oxyntomodulin and GDF-15 concentrations; (2) to investigate whether exercise-induced changes in circulating OXM and GDF-15 concentrations are correlated with subjective appetite perceptions and subsequent energy intake.

DETAILED DESCRIPTION:
Oxyntomodulin is thought to promote weight loss by suppressing appetite and energy intake and increasing energy expenditure. Acute exercise has been shown to increase the circulating concentration of satiety-related gut hormones, such as glucagon-like peptide-1 (GLP-1) and peptide YY (PYY). However, the effect of acute exercise on OXM concentrations in individuals with healthy weight has not been investigated.

GDF-15 is a cellular stress-induced cytokine which has recently been shown to suppress appetite. A few studies have explored the effect of acute exercise on GDF-15 concentrations but the findings are conflicting. Some studies have shown that acute exercise, which provides a transient physiological stress, increased GDF-15 concentrations, but other studies have not found any influence of exercise on GDF-15 concentrations. In addition, whether post-exercise appetite perceptions and subsequent energy intake are influenced by exercise-related changes in OXM or GDF-15 concentrations remains unknown.

To explore the impact of acute moderate-intensity continuous exercise on OXM and GDF-15 levels, alongside subjective appetite perceptions and subsequent energy intake, all participants in this crossover study engaged in both exercise and control trials, with a minimum one-week interval between each.

During the exercise trial, participants were asked to arrive at the lab at 8.30 am, having fasted overnight for 10 hours (except plain water). Participants were asked to rest in the lab for 30 minutes. During the resting period, a cannula was positioned in the participants' arm and a mask was fitted on the face in the last five minutes of the rest to allow for the collection of exhaled air during exercise. After the resting period, participants were asked to exercise at an intensity of 70 percent of their peak oxygen uptake for an hour before resting in the lab for a further 2.5 hours. Venous blood samples were collected before (0 minutes) and after (60, 90, 120, 150, 180, and 210 minutes) exercise and ad libitum energy intake was assessed 1 h after exercise completion. For the control trial, participants replicated all the procedures of the exercise trial except they rested for 1 h as the exercise counterpart.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.5-24.9 kg/m²;
* Habitually consume three meals a day;
* Able to run continuously for 1 hour;
* Not currently dieting and weight stable for 3 months (< 3 kg change in weight);
* No severe dislike or allergy to any of the study food;
* Regular menstrual cycle in the past 6 months.

Exclusion Criteria:

* Smokers (vaping is considered smoking in this study);
* Individuals with medical conditions (e.g., diabetes, heart condition);
* Individuals taking medications that may influence the study outcomes;
* Individuals with clinically diagnosed eating disorders.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Oxyntomodulin | Blood samples were collected for oxyntomodulin measurements at 0 (baseline), 60, 90, 120, 150, 180, 210 minutes in each trial.
  (pmol/L)
Growth Differentiation Factor 15 | Blood samples were collected for GDF-15 measurements at 0 (baseline), 60, 90, 120, 150, 180, 210 minutes in each trial.
  (pg/mL)

SECONDARY OUTCOMES:
Visual analogue score (VAS) for subjective appetite | VAS was measured at 0 (baseline), 60, 90, 120, 150, 180, 210 minutes in each trial.
  Subjective appetite sensations were assessed using 100mm visual analogue scales to measure four appetite constructs: 'hunger', 'fullness,' 'desire to eat' and 'expected food intake'.
Energy intake | Ad libitum pasta meal provided at 120 minutes.
  (kcal); participants were required to self-serve from a large bowl containing an amount of pasta in excess of expected consumption for 30 minutes and were instructed to stop eating when they reach volitional satiation. The remaining food was weighed and subtracted from the known quantity initially presented to calculate ad libitum energy intake.

CONTACTS AND LOCATIONS:
Overall Officials: David J Stensel, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available to researchers upon request.